CLINICAL TRIAL: NCT00175123
Title: Phase 4 Study of the Effect of Botulinum-A Toxin Injected in Neurogenic Overactive Bladders of Children Born With Myelomeningocele
Brief Title: Effect of Botulinum Toxin in Neurogenic Bladders in Children With Myelomeningocele
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Bettina Jorgensen, MD, Aarhus University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Botox; J.nr.2612-2319; J.nr.20030155
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Myelomeningocele; Bladder, Neurogenic
Keywords: Myelomeningocele; Neurogenic Bladder; Intervention; Botulinum A toxin; Oxybutynin
MeSH Terms: conditions — Meningomyelocele; Urinary Bladder, Neurogenic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum A toxin — Intravesical injection. 12 IE/kg b.w.

SUMMARY:
The purpose of this study is to examine how injection of botulinum toxin in the bladder affects bladder function. The trial is carried out in children born with malformation of the spinal cord and subsequent overactive bladders. The purpose of treating the bladder (with different drugs) is to prevent damage to the kidneys and renal function. The aim of this study is to compare a conventionally used drug (oxybutynin) with botulinum toxin. The hypothesis of the study is that botulinum toxin is equal to oxybutynin in the treatment of overactive bladder.

DETAILED DESCRIPTION:
Neurogenic bladder is often seen in children with myelomeningocele, tumors in the spinal canal, or a traumatized spinal cord. The majority of the patients have high pressure bladders which can lead to reflux and frequent infections in the urinary tract. Although children experience insufficient bladder emptying, many of them also experience urinary incontinence and have to perform clean intermittent catheterization (CIC). If no intervention is made, the children are at high risk of renal deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Myelomeningocele
* Neurogenic bladder with untreated leak point pressures > 40 mmH2O
* Treated with oxybutynin or other parasympatholytics

Exclusion Criteria:

* Acute urinary tract infection
* Compromised neuromuscular transmission

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-03 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Bladder capacity and pressures: measures from cystometry | at 4 weeks and 6 months

SECONDARY OUTCOMES:
Urinary continence: score from an incontinence rating scale | 2 days before and 4 weeks and 6 months after
Constipation: score on the Bristol scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jorgensen, MD, Principal Investigator — Department of Urology, Aarhus University Hospital
Locations (1):
- Department of Urology, Aarhus University Hospital, Section Skejby, Aarhus, Aarhus N, Denmark